CLINICAL TRIAL: NCT03786601
Title: High-risk HPV Infection and Vaginal Microbiota in Postmenopausal Women
Brief Title: Postmenopausal Women With Vaginal Microbiota
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, shuwang, Associate Professor, Peking Union Medical College Hospital
Other Study IDs: PMWVM
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: HPV-Related Squamous Cell Carcinoma
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A,: High-risk HPV infection in postmenopausal women
  Interventions: Other: Observation
- Group B: High-risk HPV negative in postmenopausal women
- Group C: High-risk HPV infection in gestational women
  Interventions: Other: Observation
- Group D: High-risk HPV negative in gestational women

INTERVENTIONS:
Other: Observation — The participants were assigned to different groups according to the results of HPV detection.
  Groups: Group A,; Group C

SUMMARY:
Since other genital infections enhance HIV susceptibility by inducing inflammation, the investigators study the relationship between the vaginal microbiota composition and the risk of HPV infection, cervical cytological abnormalities in postmenopausal women.

DETAILED DESCRIPTION:
Persistent infection with oncogenic Human Papillomavirus (HPV) is necessary but not sufficient for the development of cervical cancer. Additional factors correlated with HPV persistence include immunodeficiency caused by HIV, smoking, use of oral contraceptives and, more recently reported, vaginal dysbiosis. In a state of dysbiosis, there is a marked reduction of Lactobacillus and a high diversity of bacteria, with increased abundance of anaerobic bacterial species. Owing to the decrease of estrogen level and cervical atrophy in postmenopausal women, cervical cytology is more prone to abnormal changes than in premenopausal women. Clinically, cervical lesions in elderly women are easily neglected. Therefore, cervical cancer in the elderly is usually found in advanced stage, with poor prognosis and more complications of treatment. Based on this, the investigators are going to analyze the changes of microbiota in women with high-risk HPV and the cervical lesions in menopausal women. And the investigators hope to figure out the difference and change in microbiota to realize the tanning of cervical lesions.

ELIGIBILITY:
Inclusion Criteria:

* Those are aged 20 to 75 years old, have had vaginal intercourse more than 3 years, and aren't in menstrual, pregnancy or puerperium period.

Exclusion Criteria:

* Those have no vaginal intercourse, and can't cooperate the examiner. Women who are HIV or hepatitis B/C positive, have autoimmune disorders and systemic disease (like diabetes mellitus, hormone treatment diseases, severe liver and kidney dysfunction), or have severe mental illness and malignant tumors are also excluded. At the same time, all the participants should meet the following requirements: no vagina douching within last 2 days, no vaginal intercourse within last 3 days, no systemic application of antifungal agents or antibiotics or pessaries within last 14 days of sampling.

Ages: 20 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The participants sample was referred to the paper already published.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2018-12-25 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal microbiota and HR-HPV infection in menopausal women | 6 months
  The persistence vaginal organism in HPV infection menopausal women

SECONDARY OUTCOMES:
The difference of vaginal microbiota in different age groups | 6 months
  The difference of vaginal microbiota in different age groups with HR-HPV infection
The difference of vaginal microbiota in different age groups | 6 months
  The difference of vaginal microbiota in different age groups without HR-HPV

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China